CLINICAL TRIAL: NCT04568759
Title: Randomized Controlled Trial to Evaluate the Effect of a Postural Re-education Intervention Compared to Standard Care on Scoliosis Progression in Adolescent
Brief Title: Effect of a Postural Re-education Intervention Compared to Standard Care on Scoliosis Progression in Adolescent
Acronym: RCT-RPG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Laval University (Other); Shriners Hospitals for Children (Other); Université de Montréal (Other); CHU de Québec (Unknown)
Responsible Party: Principal Investigator, Carole Fortin, Associate professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-3065_RCT-RPG
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: adolescent idiopathic scoliosis; Global postural re-education; back pain; quality of life; trunk imbalance; inter muscular coherence; respiratory function; functional performance
MeSH Terms: conditions — Back Pain; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care group (Active Comparator): Observation or brace plus conventional physiotherapy exercises on video
  Interventions: Other: Global postural re-education
- GPR group (Experimental): GPR interventions added to standard care (observation or brace)
  Interventions: Other: Global postural re-education

INTERVENTIONS:
Other: Global postural re-education — GPR consists of active treatment posture and sensorimotor control exercises to regain back muscle symmetry and correct posture in daily activities

SUMMARY:
The aim of this project is to verify the effect of the global postural reeducation (GPR) intervention used in physiotherapy on scoliosis progression (scoliosis angle), back pain, quality of life, respiratory function, trunk posture and trunk muscle functioning and walking endurance. To do so, we will recruit 144 participants at three scoliosis specialized Centers. Participants will be randomly allocated to the standard of care (SC) group (observation or brace plus home video of exercises for 12 months) or to the GPR group (SC plus individual sessions once a week for 6 months and individual sessions alternating with telerehabilitation sessions once per two weeks between 6 and 12 months). At initial, 6, 12- and 24-months evaluation, participants will have x-ray, complete self-report questionnaires to document back pain and quality of life. Thereafter, measurement of trunk posture, electromyography activity of the back muscles, excursion of the diaphragm muscle using echography and respiratory function as well as distance covered using the 6-minute walk test for walking endurance will be done. We believe that GPR intervention may prevent scoliosis progression and improve physical health and quality of life in adolescence.

ELIGIBILITY:
Inclusion Criteria:

* aged between 10 and 16 years old,
* Cobb angle between 15º and 45º,
* Risser sign ≤3 (skeletal growth incomplete),
* with a risk of progression index > 1.3,
* having recent x-rays (4-6 weeks),
* ability to travel weekly to attend GPR intervention

Exclusion Criteria:

* patients with diagnosis other than AIS,
* patients who are planned for surgery,
* have had surgery,
* worn a brace for at least three months prior to GPR intervention

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Cobb angle of at least 5 degrees | 6, 12 and 24 months
  Angle measured on radiograph for scoliosis progression

SECONDARY OUTCOMES:
Back pain on the Numerical Pain Rating Scale | 6, 12 and 24 months
  Intensity of back pain on the Numerical Pain Rating Scale (0-10, where 0 indicates no pain et 10 the worst imaginable pain)
Italian Spine Youth Quality of Life questionnaire | 6, 12 and 24 months
  Quality of life: score is between 0 and 100, where 100 represents a higher quality of life
Trunk imbalance | 6 and 12 months
  The right/left horizontal deviation between the plumb line placed at C7 and S1 calculated in mm
Diaphragm excursion | 6 and 12 months
  Diaphragm excursion using ultrasound imaging in mm

CONTACTS AND LOCATIONS:
Overall Officials: Carole Fortin, PhD, Principal Investigator — CHU Sainte-Justine/Université de Montréal
Locations (2):
- Canada (2):
  - CHU Sainte-Justine, Montreal, Quebec
  - Centre interdisciplinaire de recherche en réadaptation et intégration sociale/Université Laval, Québec

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD